CLINICAL TRIAL: NCT02565316
Title: Efficacy of Nepeta Menthoides Boiss & Bohse Freeze Dried Extract on Anxiety of Patients With Depression: a Double-blind Randomized Controlled Clinical Trial
Brief Title: Efficacy of Nepeta Menthoides Extract on Anxiety of Patients With Depression: a Double-blind Randomized Controlled Clinical Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sepideh Kolouri, Shiraz University of Medical Sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9470-7440
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nepeta menthoides Boiss & Bohse freeze dried extract capsule (Active Comparator)
  Interventions: Drug: Nepeta menthoides Boiss & Bohse freeze dried extract
- Sertraline capsule (Active Comparator)
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Nepeta menthoides Boiss & Bohse freeze dried extract
  Arms: Nepeta menthoides Boiss & Bohse freeze dried extract capsule
Drug: Sertraline
  Arms: Sertraline capsule

SUMMARY:
The aim of this study is to assess the efficacy of Nepeta menthoides as an anti anxiety herbal remedy for depressed patients , in a 6 week randomized double-blind controlled trial. A total of 70 adult outpatients between 18-65 ages referring to psychiatry clinic of Shiraz medical university, who having depression according to Persian-language version of the Beck Depression Inventory-Second edition and get score above 11 according to Persian version of Beck Anxiety Inventory (BAI) and diagnosis is confirmed by at two psychiatrists are randomly allocated into two groups and assign to receive 400 mg of freeze dried powder of Nepeta menthoides or 50 mg of sertraline in the uniformed capsules twice daily (in the morning and 1-2 hours before sleeping time at night). Exclusion criteria were pregnancy and lactation, allergy to N. menthoides and Lamiaceae family, patients with suicidal thoughts or previous suicidal attempt, patients with unstable cardiac, renal and hepatic diseases, seizure and hypothyroidism and patients who used substances or alcohol and patients who had indication for electroconvulsive therapy.. Severity of anxiety (by Persian version of Beck Anxiety Inventory (BAI)) and also common possible side effects of drugs will assess in baseline, 2nd week, 4th week and then two weeks after the end of the intervention (in 6th week)

ELIGIBILITY:
Inclusion Criteria:

1. having depression according to Persian-language version of the Beck Depression Inventory-Second edition
2. get score above 7 according to Persian version of Beck Anxiety Inventory (BAI)

Exclusion Criteria:

1. pregnancy and lactation
2. allergy to N. menthoides and Lamiaceae family
3. patients with suicidal thoughts or previous suicidal attempt
4. patients with unstable cardiac, renal and hepatic diseases, seizure and hypothyroidism
5. patients who used substances or alcohol
6. patients who had indication for electroconvulsive therapy -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Persian version of Beck Anxiety Inventory (BAI) | 6 weeks

SECONDARY OUTCOMES:
side effects of intervention drugs | 6 weeks